CLINICAL TRIAL: NCT01050491
Title: Effect of a Receptor Antagonist of Endothelin 1 (Sitaxsentan, Thelin) on Bronchial Remodeling in Severe Asthma With Fixed Bronchial Obstruction
Brief Title: Study on the Effects of Sitaxsentan on Airway Remodeling in Patients With Severe Asthma
Acronym: Sitax
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sitaxentan is not commercialized anymore
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C07-25
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Effect of Sitaxsentan on Airway Remodeling in Severe Asthma
Keywords: asthma; airway remodeling; airway obstruction
MeSH Terms: conditions — Asthma; Airway Remodeling; Airway Obstruction | interventions — sitaxsentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sitaxsentan, airway remodeling (Placebo Comparator): Blinded, randomised placebo-controlled trial involving two parallel groups of severe asthmatic patients with irreversible airflow obstruction (FEV1≤ 70% of predicted) .
  Interventions: Drug: sitaxentan; Drug: placebo
- placebo, airway remodeling (Placebo Comparator): Blinded, randomised placebo-controlled trial involving two parallel groups of severe asthmatic patients with irreversible airflow obstruction (FEV1≤ 70% of predicted) .
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sitaxentan — 100 mg once a day during one year. Bronchial fibroscopy
  Arms: sitaxsentan, airway remodeling
Drug: placebo — placebo, one per day, during one year. Bronchial fibroscopy

SUMMARY:
Introduction. Despite adequate steroid therapy, a subpopulation of approximately 10% of asthmatics develops severe persistent airflow obstruction. It is now widely agreed that the latter is the consequence of a remodeling process of the airways, characterized by an increase in airway smooth muscle mass, mucus gland hypertrophy, increased thickness of the subepithelial basement membrane, extracellular matrix protein deposition, angiogenesis, fibroblast and myofibroblast accumulation. These phenomena are responsible for airway wall thickening and for decreased airway caliber leading to persistent airflow obstruction.

Endothelin-1 (ET-1) is a small peptide, synthesized in the lung by airway epithelial and smooth muscle cells, as well as inflammatory cells. ET-1 induces bronchoconstriction, mediates eosinophils recruitment during allergic inflammation and contributes to airway remodeling by inducing fibroblasts and smooth muscle cells differentiation and proliferation. In a recent work from Inserm Unit 700, it has been shown that ET-1 was overexpressed in epithelial cells from severe asthmatic patients as compared to patients with less severe disease, and that ET-1 expression was strongly correlated with airway obstruction (measured by FEV1) and on bronchial biopsies with airway smooth muscle areas. In another study, we have shown that a polymorphism of the receptor for ET-1 was strongly associated with the degree of airway obstruction in a population of asthmatic patients. All these data suggest that inhibition of the ET-1 pathway could be a potential therapeutic option in patients with steroids refractory asthma and irreversible airway obstruction. Bosentan, a specific inhibitor of ET-1 receptors which is actually used in patients with pulmonary hypertension, improves survival and inhibits vascular remodeling.

Aim and strategy. To study the impact on airway remodeling and clinical status of an antagonist of the endothelin receptors (Sitaxentan 100mg/day) over a 12-month period, in a prospective randomised placebo-controlled trial involving two parallel groups of 25 severe asthmatic patients with irreversible airflow obstruction (FEV1≤ 70% of predicted) . Various hallmarks of airway remodeling will be analyzed on bronchial biopsy specimens by immunohistochemistry and morphometry. These findings will be correlated with the results of pulmonary function tests. Twenty-five patients will be included in each group. Remodeling will be measured on bronchial biopsies performed during fiberoptic bronchoscopy at inclusion and after one year, by assessing smooth muscle area, submucosal fibroblasts count and basement membrane thickness. Every 3 months, bronchial obstruction (FEV1), clinical status, asthma exacerbations, steroids use, need for emergency care, asthma symptoms and quality of life will be assessed. Evaluation of airway inflammation will be assessed every 3 months by exhaled NO and induced sputum cytology.

This proof of concept study will validate ET-1 as a new molecular target for treating airway remodeling in patients with severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* 50 non smoking (25 on active treatment and 25 on placebo) patients with severe asthmatic patients (age over 18 and less than 70) and irreversible airflow obstruction (FEV1≤ 70% of predicted)

Exclusion Criteria:

* Abnormal liver chemistry at inclusion, female without acceptable contraceptive methods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in airway remodeling analyzed on bronchial biopsy specimens at inclusion and after one year by immunohistochemistry and morphometry (smooth muscle area, and submucosal fibroblasts count). | 2 years

SECONDARY OUTCOMES:
FEV1,clinical status, asthma exacerbations, steroids use, need for emergency care, asthma symptoms and quality of life,exhaled NO and induced sputum cytology. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Investigation center 07, Hopital Bichat, Paris, France